CLINICAL TRIAL: NCT03383588
Title: Efficacy of Subcutaneous Infiltration With Local Anesthetic During Elective Cesarean Delivery for Postoperative Pain Control: a Randomized Controlled Trial
Brief Title: Subcutaneous Bupivacaine Decrease Post-op Pain in Patients Undergoing C-Section
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: study was published during initial recruitment that showed no difference
Sponsor: Montefiore Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Supportive Care
Other Study IDs: 2017-8094
Record Dates: First submitted 2017-12-14; First posted 2017-12-26 (Actual); Results first posted 2020-01-13 (Actual); Last update posted 2020-01-13 (Actual); Status verified 2019-12

CONDITIONS: Pain, Referred
MeSH Terms: conditions — Pain, Referred | interventions — Bupivacaine; Morphine; Fentanyl; Analgesics, Opioid; Epinephrine; Saline Solution; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (3):
- bupivacaine 0.25% (Active Comparator): standard intrathecal bupivacaine (Marcaine) 0.75% 1.5-1.7 ml, intrathecal morphine (Duramorph) 150mcg plus intrathecal fentanyl 10 mcg + 20 ml subcutaneous bupivacaine (Marcaine) 0.25%
  Interventions: Drug: Bupivacaine; Drug: Morphine; Drug: Fentanyl
- bupivacaine 0.25% + epinephrine (Active Comparator): standard intrathecal bupivacaine (Marcaine) 0.75% 1.5-1.7 ml, intrathecal morphine (Duramorph) 150mcg plus intrathecal fentanyl 10 mcg + 20 ml subcutaneous bupivacaine (Marcaine) 0.25% with Epinephrine
  Interventions: Drug: Bupivacaine; Drug: Morphine; Drug: Fentanyl; Drug: Epinephrine
- Saline Solution (Placebo Comparator): standard intrathecal bupivacaine (Marcaine) 0.75% 1.5-1.7 ml, intrathecal morphine (Duramorph) 150mcg plus intrathecal fentanyl 10 mcg + 20 ml subcutaneous NACL 0.9% (placebo)
  Interventions: Drug: Bupivacaine; Drug: Morphine; Drug: Fentanyl; Other: Saline solution

INTERVENTIONS:
Drug: Bupivacaine — 20 ml subcutaneous bupivacaine (Marcaine) 0.25%. Bupivacaine is an anesthetic which can numb an area of the body to relieve pain during surgery or medical procedures, childbirth, and dental work.
  Other Names: Marcaine
Drug: Morphine — intrathecal morphine (Duramorph) 150mcg. DURAMORPH (morphine injection) is a systemic narcotic analgesic for administration by the intravenous, epidural or intrathecal routes. It is used for the management of pain not responsive to non-narcotic analgesics. DURAMORPH (morphine injection) administered epidurally or intrathecally, provides pain relief for extended periods without attendant loss of motor, sensory or sympathetic function.
  Other Names: Duramorph
Drug: Fentanyl — intrathecal fentanyl 10 mcg. Fentanyl (also spelled fentanil) is an opioid which is used as a pain medication and together with other medications for anesthesia.
  Other Names: Opioid
Drug: Epinephrine — Epinephrine injection is used along with emergency medical treatment to treat life-threatening allergic reactions caused by insect bites or stings, foods, medications, latex, and other causes. Epinephrine is in a class of medications called alpha- and beta-adrenergic agonists (sympathomimetic agents). It works by relaxing the muscles in the airways and tightening the blood vessels.
  Other Names: Adrenaline
  Arms: bupivacaine 0.25% + epinephrine
Other: Saline solution — 20 ml subcutaneous NACL 0.9% - saline solution is the placebo
  Other Names: Sodium Chloride
  Arms: Saline Solution

SUMMARY:
The purpose of this study is to determine if giving an injection of numbing medication at the incision at the end of cesarean will help control pain AFTER cesarean delivery. This study seeks to assess pain relief with incisional infiltration of local anesthetic during cesareans performed under spinal anesthesia also using intrathecal opioids. Participants will receive the usual regimen of pain medication in spinal anesthesia. At the end of the cesarean delivery, while the participants are still under the spinal medication, participants will receive an injection, at the incision, either numbing medication (with or without epinephrine) or sterile saline. After the cesarean delivery, participants will receive, by mouth, commonly prescribed pain medications - these medications are oxycodone (an opioid/ narcotic), acetaminophen (or more commonly known as Tylenol), and ibuprofen.

DETAILED DESCRIPTION:
The study assesses addition of subcutaneous bupivacaine with and without epinephrine to the standard intrathecal morphine/fentanyl combination given during spinal anesthesia during elective cesarean delivery on postoperative pain control as measured by postoperative usage of oral opioids and a postoperative pain assessment scale. Comparing post-op pain scores and oxycodone usage in patients who receive just intrathecal morphine to patients who receive intrathecal morphine plus subcutaneous bupivacaine .25%, to patients who receive bupivacaine .25% with epinephrine 1:200,000.

After cesarean delivery, all groups will actively control the use of post-operative pain medication by indicating to the care nurse whether or not pain medication is desired. Pain control for all groups will be the standard pain treatment: ibuprofen for mild to moderate pain and percocet (oxycodone) for severe pain.

The U.S. Food and Drug Administration (FDA) has approved bupivicaine as an anesthetic and for pain but the FDA has not approved bupivicaine to be given specifically for postoperative cesarean pain. Acetaminophen, oxycodone and ibuprofen are being used as part of routine clinical care for pain control after cesarean. Fentanyl and duramorph are being used in spinal anesthesia and are FDA approved for regional anesthesia and used for this purpose in routine clinical care.

ELIGIBILITY:
Inclusion criteria:

* elective cesarean delivery
* planned spinal anesthesia

Exclusion criteria:

* Non-English speaking
* Urgent or emergent cesarean delivery
* Active labor [defined as: >4cm cervical dilation or regular contractions noted on tocometer (>2 contractions in a 10 minute period for 30 consecutive minutes)]
* Chronic antepartum opioid use
* History of substance abuse (alcohol or drug)
* Current tobacco use
* Chronic steroid use

Ages: 17 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Gender Based: Yes — Pregnant women undergoing Cesarean Section under spinal anesthesia
Enrollment: 26 (Actual)
Dates: Start 2018-07-19 (Actual); Primary Completion 2018-08-17 (Actual); Study Completion 2018-12-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jeffrey Bernstein, MD, Principal Investigator — Montefiore Medical Center
Locations (1):
- Albert Einstein College of Medicine/ Montefiore Medical Center, The Bronx, New York, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Bupivacaine 0.25% | Bupivacaine 0.25% + Epinephrine | Saline Solution
Started | 8 | 9 | 9
Completed | 8 | 9 | 9
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: baseline population presenting for scheduled c-section; study terminated early secondary to other similar published study showing no difference
Groups:
- Total: Total of all reporting groups
Arm/Group | Bupivacaine 0.25% | Bupivacaine 0.25% + Epinephrine | Saline Solution | Total
Number analyzed (Participants) | 8 | 9 | 9 | 26
Age, Continuous [Mean (Full Range); unit: years] | 29 [23 to 35] | 34 [28 to 40] | 29 [27 to 37] | 31 [23 to 40]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8 | 9 | 9 | 26
  Male | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 1 | 1 | 1 | 3
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 0 | 1 | 3 | 4
  White | 1 | 1 | 0 | 2
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 6 | 6 | 5 | 17
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 8 | 9 | 9 | 26
Estimated Blood Loss (EBL) [Mean (Full Range); unit: ml of blood] | 900 [400 to 2000] | 855 [500 to 1200] | 744 [600 to 1200] | 830 [400 to 2000]

OUTCOME MEASURES:

1. Primary Outcome: Amount of Supplemental Oxycodone Used
Description: Cumulative opioid pain medication used in the first 24 hours postoperatively as recorded in the medical record
Time Frame: 4-24 hours post operative
Population: all patients
Measure: Mean (Full Range); unit: mg of supplemental oxycodone
Arm/Group | Bupivacaine 0.25% | Bupivacaine 0.25% + Epinephrine | Saline Solution
Number analyzed (Participants) | 8 | 9 | 9
mg of supplemental oxycodone | 19 [10 to 30] | 25 [15 to 40] | 23 [10 to 40]

ADVERSE EVENTS:
Time Frame: The participants were followed for a period of 6 months after initial date of recruitment for adverse events via medical record review
Description: Does not differ
Arm/Group | Bupivacaine 0.25% | Bupivacaine 0.25% + Epinephrine | Saline Solution
All-Cause Mortality (participants affected / at risk) | 0/8 | 0/9 | 0/9
Serious Adverse Events (participants affected / at risk) | 1/8 | 2/9 | 2/9
Other Adverse Events (participants affected / at risk) | 0/8 | 0/9 | 0/9
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Bupivacaine 0.25% (N=8) | Bupivacaine 0.25% + Epinephrine (N=9) | Saline Solution (N=9)
Large intraoperative blood loss (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 0 (0) | 1 (1) — Patient had preoperative anemia and a large intraoperative blood loss secondary to dense intraabdominal adhesions requiring 2 units pRBC's
Postpartum re-admission to hospital (not OBGYN related) (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0) — Patient was admitted to general surgery service 1 month postpartum for acute cholecystitis requiring a cholecystectomy
Large intraoperative blood loss (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 1 (1) | 0 (0) — Patient had a placenta previa that was adhered to the lower intrauterine segment intraoperatively, had a large intraoperative blood loss not requiring transfusion, and had a uterine tamponade balloon placed intraoperatively
Postpartum readmission to hospital (OBGYN related) (Pregnancy, puerperium and perinatal conditions) | 1 (1) | 0 (0) | 0 (0) — Patient was admitted one week postoperatively for severe postpartum preeclampsia
Large intraoperative blood loss (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 0 (0) | 1 (1) — Patient had a placenta previa that was adhered to the lower intrauterine segment intraoperatively, had a large intraoperative blood loss not requiring transfusion, and had a uterine tamponade balloon placed intraoperatively

LIMITATIONS AND CAVEATS:
Early termination leading to small numbers of subjects and Technical problems with measurement leading to unreliable or uninterpretable data; Study terminated early secondary to similar study published showing no difference in outcomes

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Informed Consent Form (2018-05-18): https://cdn.clinicaltrials.gov/large-docs/88/NCT03383588/ICF_000.pdf
  • Study Protocol and Statistical Analysis Plan (2018-07-11): https://cdn.clinicaltrials.gov/large-docs/88/NCT03383588/Prot_SAP_001.pdf